CLINICAL TRIAL: NCT03659708
Title: Prospective Multicentre Randomized Clinical Trial on the Management of Pregnancies With High Risk of Venous Thrombosis
Brief Title: Pregnancy and Risk of Venous Thromboembolism
Acronym: PRESCOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL18_0032; 2018-A02777-48 (Other: ID-RCB)
Record Dates: First submitted 2018-08-13; First posted 2018-09-06 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Thromboembolism; Pregnancy
Keywords: low molecular weight heparin (LMWH); Lyon VTE-score; pregnancy; thromboprophylaxis; venous thromboembolism; quality of life; cost utility
MeSH Terms: conditions — Thromboembolism; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lyon-VTE score (Experimental): 300 adult pregnant women with a personal history of VTE and/or known thrombophilia, will be randomly included in this group and their VTE risk during pregnancy will be managed according to the Lyon-VTE score :
  The Lyon score classifies patients into 3 risk categories and directs the preventive LMWH prescription:
  * A score strictly less than 3 indicates a moderate thrombotic risk: the patient does not receive LMWH in ante-partum;
  * A score between 3 and 5 indicates a high thrombotic risk: a preventive dose LMWH is introduced in the third trimester (from the beginning of the 7th month);
  * A score greater than or equal to 6 indicates a very high thrombotic risk: LMWH at a preventive dose is prescribed throughout the ante-partum.
  All patients receive an elasto-compression prescription and daily physical activity is recommended throughout pregnancy (except obstetric contraindication).
  All patients also receive systematic preventive LMWH treatment postpartum for 6 weeks.
  Interventions: Procedure: Lyon-VTE score
- recommendations currently available (Experimental): 300 adult pregnant women with a personal history of VTE and/or known thrombophilia, will be randomly included in this group and their VTE risk during pregnancy will be managed according to the last ACCP guidelines or UK guidelines or Canadian recommendations or French recommendations, according to the habits of the center.
  Interventions: Procedure: recommendations currently available

INTERVENTIONS:
Procedure: Lyon-VTE score — follow-up at 3 months, 5 months, 7 months during pregnancy and 3 months and 12 months after delivery.
  Arms: Lyon-VTE score
Procedure: recommendations currently available — follow-up at 7 months during pregnancy and 3 months and 12 months after delivery.
  Arms: recommendations currently available

SUMMARY:
The management of venous thromboembolism (VTE) risk in pregnancy still remains a challenge. An individual assessment of the VTE risk is crucial for optimal thromboprophylaxis, but there is no validated tool to help clinicians stratify the risk in pregnant women and introduce prophylactic anticoagulation at the appropriate time. Recommendations mostly based on case-control studies and expert opinions do not accurately reflect the physician's need. In view of the lack of international recommendations with a high level of evidence regarding prophylactic treatment of pregnant women at risk of thrombosis, the use of a risk stratification tool that takes all individual risk factors for VTE into consideration and which aids decisions over prophylaxis regimens may help. Investigators have previously described a VTE risk score (the Lyon-VTE-score), rating patients at increased risk of VTE and recommending individually tailored management. A retrospective evaluation of the initial score showed favorable outcomes in pregnancies with a high risk of thrombosis. A subsequent multicenter prospective study reported promising results using this score and related management strategy. The efficacy and safety after 10 years of prospective use of the Lyon-VTE-score in daily practice to guide the prescription of antithrombotic prophylaxis during pregnancy was recently evaluated and the results showed that the Lyon-VTE-score allows a standardized approach with objective criteria and can help non-specialized centers and young doctors manage these high-risk pregnancies.

The results of previous studies provide consistent conclusions on the safety and efficacy of the approach of investigators and give background for a medico-economic study to evaluate costs and consequences of this procedure. The most recent study (2005) evaluating the cost of prophylaxis in pregnant women, evaluated this cost as $1292 for each 6-week cycle of treatment. In addition, the use of such a score offers the prospect of personalized medicine, which is probably more cost-efficient compared to "inclusive, equal treatment for all".

In antepartum, the decision to administer thromboprophylaxis should be considered on an individual basis with regard to lowering the absolute risk of thrombosis, the inconvenience of daily subcutaneous heparin therapy and the potential risks of bleeding, heparin-induced thrombocytopenia and osteoporosis. An individual assessment of the VTE risk is crucial for optimal thromboprophylaxis, but there is no validated tool to help clinicians to stratify VTE risk in pregnant women and to introduce prophylactic anticoagulation at the right time.

Most of the recommendations are grade 2C. They are mostly based on case-control studies and expert opinions and do not entirely highlight the physicians' need. The originality of this approach is the use of a risk stratification tool that takes all individual risk factors for VTE into consideration and that aids the decision-making process of antenatal anti-thrombotic prophylaxis. This study will personalize care using a score to individually assess the risk and propose appropriate prevention.

The main objective of this study is to conduct a medico-economic study to evaluate the efficiency of an innovative strategy integrating the Lyon-VTE-score in the management of pregnant patients with venous thromboembolism risk versus standard care.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant women at high risk of VTE (with a personal history of VTE and/or thrombophilia)
* giving informed consent to participate to the study

Exclusion Criteria:

* contraindication to heparin therapy,
* women with obstetrical complications only, with no history of VTE (pre-eclampsia, HELLP[ Hemolysis, Elevated Liver enzymes, Low Platelet count],intra-uterine growth retardation, miscarriage, etc),
* patients with a history of superficial venous thrombosis, and those with the highest VTE risk for whom clear recommendations with a high level of evidence are available (patients on long-term anticoagulants, or those with antiphospholipid syndrome or antithrombin deficiency).
* Patient participating in an ongoing study that could interfere with the study,
* Patient under legal protection measure.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2026-10-22 (Estimated); Study Completion 2026-10-22 (Estimated)

PRIMARY OUTCOMES:
cost-utility ratio | until 12 months after delivery
  Medico-economical data related to the score-based management strategy will be collected during all pregnancy and at months 3 and 12 in the postpartum period.

SECONDARY OUTCOMES:
occurrence of venous thromboembolism | until 12 months after delivery
  efficacy data related to the score-based management strategy will be collected during all pregnancy and at months 3 and 12 in the postpartum period
occurrence of bleeding complications | until 12 months after delivery
  safety data related to the score-based management strategy will be collected during all pregnancy and at months 3 and 12 in the postpartum period
Evaluation of quality of life of pregnant women at high risk of thrombosis by the EQ-5D-3L survey | until 12 months after delivery
  quality of life data will be collected during all pregnancy and at months 3 and 12 in the postpartum period using the EQ-5D-3L survey

CONTACTS AND LOCATIONS:
Overall Officials: Yesim DARGAUD, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Cardiologique L. Pradel, Bron, France

REFERENCES:
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986